CLINICAL TRIAL: NCT05543395
Title: The Reporting of Domestic Violence by Patients in the Emergency Department of the Reims University Hospital Center
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO21001
Record Dates: First submitted 2021-08-03; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Domestic Violence
Keywords: Domestic violence; Report of domestic violence; Reims University Hospital Center; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The group accepting to report
  Interventions: Behavioral: Domestic Violence Questionnaire
- The group refusing to report
  Interventions: Behavioral: Domestic Violence Questionnaire

INTERVENTIONS:
Behavioral: Domestic Violence Questionnaire — Domestic Violence Questionnaire

SUMMARY:
Domestic violence is defined as violence carried out by one of the partners in a relationship of domination. This can be verbal, psychological, physical or sexual.

Domestic violence is a real public health problem for which emergencies are at the forefront.

In this context, the emergency department of the Reims University Hospital Center, the Public Prosecutor and the association LE MARS France Victim 51 decided to set up a report on July 01, 2020.

The report consists of retrieving the identity and information relating to the violence suffered through a survey, or report card . The report card, as well as an initial certificate without the total incapacity for work written by the doctor during the consultation, will be sent immediately by secure email to the public prosecutor and the police. The emails will be processed in real time by the prosecutor on duty. The contact details with the family name, first name and telephone number will be sent to the association LE MARS France Victime 51. Reporting therefore allows the prosecutor to decide whether or not to open a criminal investigation., At the same time, this will allow us to provide support through the association providing assistance to victims of domestic violence.

The objective of this study is to describe the proportion of patients accepting to report to the public prosecutor among the patients consulting the emergency department of the Reims University Hospital Center and for whom domestic violence is known or suspected. The secondary objectives will be to describe the number of patients who are victims of proven or suspected domestic violence consulting the emergency department, as well as to describe the factors associated with the acceptance of the report.

Participation in the study will consist of completing a questionnaire specific to the study. The estimated time to complete this questionnaire is 5 minutes.

This study will allow us to know the prevalence of acceptance of the report card in the emergency department of the Reims University Hospital Center. This information will tell us if this new procedure could be beneficial for the management of domestic violence and if the majority of patients are in favor of it.

DETAILED DESCRIPTION:
I. Medical background :

Domestic violence is defined as violence carried out by one of the partners in a relationship of domination. This can be verbal, psychological, physical or sexual.

This type of violence is a real public health problem. According to a study carried out by the French government in 2018, 213 000 women aged 18 to 75 were victims of physical and / or sexual violence committed by their spouse or ex-spouse in 2018. According to this same study, 121 women and 28 men were killed by their partner or ex-partner. These figures are increasing every year, and the screening of these patients is a major issue.

A doctor is on the front line in screening for this violence. In fact, 3 to 4 women out of 10 in doctors' waiting rooms are victims of domestic violence; and one in five victims first saw a doctor after an incident. A French study carried out in 2002 also showed that 35% of consultations in an emergency department with a woman patient were related to domestic violence.

The High Authority of Health systematically recommends asking each patient and each suspicion of violence within the couple the question "are you a victim of domestic violence?". However, this recommendation remains largely insufficient as well as the assistance provided to the victims. Furthermore, only 19% of these victims say they have filed a complaint with an authority according to the High Authority of Health. Screening remains the first step in the care and identification of victims, but more measures are needed to be put in place to help these patients take legal action and get out of this vicious circle of domestic violence.

The emergencies are therefore one of the first recourse for patients who are victims of domestic violence and it is the role of the emergency physician to take all possible means to detect, help and support these victims.

In this context, the emergency department of the Reims University Hospital Center, the Public Prosecutor and the association LE MARS France Victim 51 decided to set up a report on July 01, 2020.

The report consists of retrieving the identity and information relating to the violence suffered through a survey, or report card . The report card, as well as an initial certificate without the total incapacity for work written by the doctor during the consultation, will be sent immediately by secure email to the public prosecutor and the police. The emails will be processed in real time by the prosecutor on duty. The contact details with the family name, first name and telephone number will be sent to the association LE MARS France Victime 51. Reporting therefore allows the prosecutor to decide whether or not to open a criminal investigation., At the same time, this will allow us to provide support through the association providing assistance to victims of domestic violence.

II. Goals:

The objective of this study is to describe the proportion of patients accepting to report to the public prosecutor among the patients consulting the emergency department of the Reims university hospital center and for whom domestic violence is known or suspected. The secondary objectives will be to describe the number of patients who are victims of proven or suspected domestic violence consulting the emergency department, as well as to describe the factors associated with the acceptance of the report card.

III. Investigation plan:

a. Evaluation criteria: A questionnaire composed of two parts was drawn up as part of this study. The first part will be completed by the patients thmselves and will collect information about them relating to their current circumstances and history. The second part is completed by the doctor specifying whether or not the patient has accepted to complete the report, the examinations carried out in the emergency room as well as the entry and exit diagnoses.

The main endpoint is acceptance of direct reporting to the public prosecutor. Secondary endpoints are the factors potentially associated with whether or not patients accept direct reporting to the public prosecutor.

IV. Methodology:

1. Experimental design:

   This is a cross-sectional, observational, prospective inclusion, single-center (Reims University Hospital Center) study over a period of 6 months.
2. Investigation plan:

   Participation in the study will be offered to all patients consulting the emergency reception service of the Reims University Hospital Center during the inclusion phase of the study and for whom domestic violence is proven or suspected during the interview. Information on the objectives and methods of the study will be given to them with the help of the information note. If the patient agrees to participate in the study, they will be included in the study. Participation in the study will not affect the patient's medical management.

   Participation in the study will lead to:
   * Completion of a questionnaire by the patient (on proven or suspected domestic violence)
   * A collection of data concerning the patient and their consultation at the emergency reception service.
3. Estimated recruitment time The recruitment period will be 6 months.
4. Duration of participation by subject The duration of patient participation is ad hoc, the time to complete the questionnaire, the duration of which is estimated to be 5 minutes.

V. Statistical analysis:

The data will be described using means ± standard deviation for quantitative and numerical variables and percentages for qualitative variables.

The factors associated with the acceptance of direct reporting to the public prosecutor will be sought by univariate analysis (Student's, Wilcoxon, Chi2 or Fisher's exact tests, depending on the conditions of application) and then multivariate (logistic regression).

The significance level adopted is 0.05. The data will be entered in an Epi info database (version 3.5.4). The statistical analyzes will be carried out using Epi info (version 3.5.4) and SAS (version 9.4) software, with the help of the Methodological Aid Unit of the Reims University Hospital Center.

ELIGIBILITY:
inclusion criteria:

* Adults over 18 years old
* Accepting participation in the study
* For whom domestic violence is known or suspected during the interview with the emergency doctor

exclusion criteria:

* Minors under the age of 18
* Unable to agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient, who consults in the emergency department of the Reims University Hospital Center, for whom domestic violence is known or suspected, accepting or not to report to the public prosecutor. Patient is able to agree of their own accord to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
acceptance of direct reporting to the public prosecutor | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France